CLINICAL TRIAL: NCT07113340
Title: Carina™ Platform - A Single-arm Study for Gastrectomy
Brief Title: Carina™ Surgical Platform for Minimal Radical Gastrectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, zhouyanbing, Professor, The Affiliated Hospital of Qingdao University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: China-made surgical robot 01
Record Dates: First submitted 2025-06-14; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Robotic Gastrectomy; Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- robot group (Experimental): Carina™ Surgical Platform, developed by Ronovo Surgical, Inc
  Interventions: Device: Carina™ Surgical Platform, developed by Ronovo Surgical, Inc

INTERVENTIONS:
Device: Carina™ Surgical Platform, developed by Ronovo Surgical, Inc — A modular surgical robot that offers greater flexibility in the number of instrument arms and surgical layout options.

SUMMARY:
To evaluate the safety and effectiveness of the laparoscopic surgical system（Carina™ Surgical Platform, developed by Ronovo Surgical, Inc) for use in gastrectomy.

DETAILED DESCRIPTION:
Source data verification: Cross-check between paper and electronic case report forms.

Standard Operating Procedures: The investigator is responsible for patient recruitment, while a independent statistician handles data collection and management. When source data is modified, changes must be traceable in both the electronic system and paper documents.

Statistical analysis plan: Categorical variables were analyzed using chi-square tests, while ordinal data were assessed using non-parametric tests. Continuous variables were analyzed using independent samples t-tests or non-parametric methods, as appropriate.

Handling of Missing Data: Missing data will be handled according to the classification of each dataset. For the Full Analysis Set (FAS), missing values for primary efficacy and safety endpoints will be imputed using the Worst Observation Carry Forward (WOCF) method, and considered as treatment failure or the occurrence of serious complications. No imputation will be performed for missing values in other datasets or for other secondary/exploratory endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years, any gender
* Patients with gastric cancer planned to undergo laparoscopic surgery assisted by the laparoscopic surgical system
* Agree to participate in this study and voluntarily sign the informed consent form
* Willing to cooperate with study follow-up and related examinations

Exclusion Criteria:

* BMI < 18.5 kg/m² or BMI ≥ 30 kg/m²
* Patients with severe cardiovascular diseases who cannot tolerate laparoscopic surgery
* Patients with severe respiratory diseases who cannot tolerate laparoscopic surgery
* Patients with severe coagulation disorders who cannot tolerate laparoscopic surgery
* Patients with a history of abdominal or pelvic surgery, radiotherapy, or chemotherapy who are not suitable for laparoscopic surgery
* Pregnant or breastfeeding women
* Patients currently participating in other drug or medical device clinical trials
* Patients deemed unsuitable for participation in this study by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Complications | From the beginning of surgery until hospital discharge, up to 16 weeks
  Any deviation from the expected postoperative recovery was considered an adverse event and was classified according to the Clavien-Dindo complication grading system. Only complications of grade III or above were included in the analysis.
Rate of No Surgical Conversion | From the start of surgery to the end of surgery, up to 5 hours
  No intraoperative conversion occurred from the robotic laparoscopic endoscopic surgical system-assisted procedure to another surgical instrument control system, conventional laparoscopy, or open surgery. The laparoscopic endoscopic surgical system is a medical device intended to assist the surgeon in accomplishing predefined surgical tasks. Completion of the remaining surgical procedures via laparoscopy or open surgery after the intended tasks have been performed using the system is not regarded as a conversion.

SECONDARY OUTCOMES:
Instrument Defects | From the start of surgery to the end of surgery
  Refers to unreasonable risks to human health or life posed by the surgical instruments used with the laparoscopic endoscopic surgical system during the clinical trial, under conditions of intended use. Such risks may arise from labeling errors, quality defects, malfunctions, or other device-related issues.
Incidence of Device-Related Adverse Events and Serious Adverse Events | From the beginning of surgery until hospital discharge, up to 16 weeks
  Any deviation from the expected postoperative recovery caused by surgical instruments was considered an adverse event and was classified according to the Clavien-Dindo complication grading system. Only complications of grade III or above were included in the analysis.
Postoperative Mortality Rate | Perioperative
  Postoperative death is defined as death resulting from causes directly related to the current surgical intervention.
Incidence of Postoperative Complications | From the beginning of surgery until hospital discharge, up to 16 weeks
  Any adverse event representing a deviation from the expected postoperative recovery was assessed and classified using the Clavien-Dindo complication grading system.
Pain Score | Pain assessments were performed twice: once at 24 hours after surgery and once prior to hospital discharge.
  Pain was assessed using the revised Wong-Baker FACES Pain Rating Scale, with scores ranging from 0 (no pain) to 10 (worst possible pain), indicating increasing severity.
Intraoperative Physiological Load Assessment of the Surgeon | An assessment was conducted immediately upon completion of the surgical procedure.
  Regional assessments were performed, covering the following areas: four fingers (excluding the thumb) of both hands, bilateral thumbs, bilateral dorsum of hands, wrists, forearms, upper arms, as well as the neck and back. Each region was scored on a scale from 0 to 10, with 0 indicating no discomfort and 10 indicating extreme discomfort in that specific area. Refer to: Lukasz F, Christopher S, Adrian Z, et al. Robot-assisted single-site compared with laparoscopic single-incision cholecystectomy for benign gallbladder disease: protocol for a randomized controlled trial[J]. BMC Surg. 2017 Feb 9;17(1):13.
Incidence of System Repairable Failures | An assessment was conducted immediately upon completion of the surgical procedure.
  A System Repairable Failures is defined as a malfunction occurring during robot-assisted surgery that can be resolved within a short period (within 1 hour) without causing significant disruption to the surgical workflow or alteration of the surgical procedure.
Postoperative Length of Hospital Stay | Perioperative
  Postoperative length of hospital stay was calculated as the number of days between the date of surgery and the date of discharge.
Robot-Assisted Surgery Time | During surgery
  Robot-assisted operative time was defined as the duration from the moment the surgeon initiated control of the surgical instruments to the moment the first robotic arm of the laparoscopic endoscopic surgical system was disengaged from the trocar and instrument control was concluded.
Intraoperative Transfusion Rate | During surgery
  The proportion of participants who underwent blood transfusion during the surgical procedure.
Intraoperative Mental Workload Assessment of the Surgeon | An assessment was conducted immediately upon completion of the surgical procedure.
  According to "Subjective Mental Effort Questionnaire". Refer to "van der Schatte Olivier RH, Van't Hullenaar CD, Ruurda JP, Broeders IA. Ergonomics, user comfort, and performance in standard and robot-assisted laparoscopic surgery. Surg Endosc. 2009;23(6):1365-1371. doi: 10.1007/s00464-008-0184-6." 0 is "no effort at all" and 150 is "exceptional amount of effort; "
Intraoperative Blood Loss | During surgery
  Blood loss was estimated using visual assessment, measurement via vacuum suction devices, or by weighing blood-soaked gauze.
System Setup Time | During surgery
  System preparation time was defined as the interval between the moment the first robotic arm of the laparoscopic endoscopic surgical system was docked to the trocar and the moment the surgeon gained control of the instruments to initiate the procedure.
  System preparation time was defined as the interval between the moment the first robotic arm of the laparoscopic endoscopic surgical system was docked to the trocar and the moment the surgeon gained control of the instruments to initiate the procedure.
  System preparation time was defined as the interval between the moment the first robotic arm of the laparoscopic endoscopic surgical system was docked to the trocar and the moment the surgeon gained control of the instruments to initiate the procedure.
Incidence of System Serious Failures | During surgery
  A serious system failure is defined as a malfunction occurring during robot-assisted surgery that either cannot be resolved within a short period (within 1 hour), or has a substantial impact on the surgical procedure or intraoperative workflow.
Instrument Performance Evaluation | An assessment was conducted immediately upon completion of the surgical procedure.
  The laparoscopic camera system and intraoperative surgical instruments-including the ultrasonic scalpel, electrosurgical scissors, needle holder, and grasping forceps-were evaluated on a four-grade scale: excellent, good, fair, and poor. Evaluation parameters included clarity of the surgical field, 3D visual fatigue, instrument stability, response latency, and operational flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Zhou, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- the Affiliated Hospital of QIngdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Investigators will not share IPD unless contact the study responsible party and obtain consent.